CLINICAL TRIAL: NCT07402382
Title: Effects of an Amylopectin Chromium Blend on Whole-Body Protein Kinetics and Glucose Control in Peri/Post-Menopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrition 21, Inc. (Industry)
Collaborators: The Center for Applied Health Sciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EH-01-2025
Record Dates: First submitted 2025-10-22; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Glucose Monitoring, Continuous; Whole Body Protein Metabolism; Peri-menopausal Women; Post-menopause
Keywords: Glucose; protein metabolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- Active 1 (Experimental): Standard dose
  Interventions: Dietary Supplement: Amylopectin-chromium blend
- Active 2 (Experimental): Concentrated dose
  Interventions: Dietary Supplement: Amylopectin-chromium blend

INTERVENTIONS:
Dietary Supplement: Amylopectin-chromium blend — Amylopectin-chromium blend, 2 g
  Arms: Active 1
Dietary Supplement: Amylopectin-chromium blend — Amylopectin-chromium blend in a concentrated format (100 mg)
  Arms: Active 2
Dietary Supplement: Placebo — Amylopectin, 2 g
  Arms: Placebo

SUMMARY:
The goal of this study is to better understand how an amylopectin chromium blend may influence whole body protein balance in women during midlife, when hormonal changes can adversely affect protein metabolism and muscle maintenance. Continuous glucose monitoring will also be used to assess glycemic control over a 24-hour period.

The main questions the study aims to answer are:

* Does the use of an amylopectin chromium blend in peri- and post-menopausal women help to support positive protein balance
* Can the affect be achieved using a concentrated dose

Researchers will compare the nutritional supplement to a placebo (amylopectin alone) to see if the amylopectin chromium blend can promote positive protein balance. A concentrated dose of the supplement will also be evaluated for comparative effectiveness.

Participants will:

* Consume the nutritional supplement (standard or concentrated dose) or placebo acutely after a short resistance exercise bout
* Complete four in-person visits, including the single-day intervention

Results from this research may help guide future nutritional strategies to support healthy aging, muscle function, and overall metabolic health.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled clinical trial will evaluate the effects of two dosage forms of an amylopectin-chromium blend on whole-body protein balance in peri- and post-menopausal women. The study will employ a stable isotope tracer methodology to quantify acute changes in protein synthesis and breakdown following a standardized resistance exercise bout and protein ingestion. Continuous glucose monitoring will assess the impact of the supplement on glycemic control over a 24-hour period.

Approximately 60 apparently healthy women, aged 40-65 years, will be enrolled at a single clinical site (The Center for Applied Health Sciences, Canfield, OH). Participants will complete four in-person visits over a 2-3-week period: one screening visit and three testing visits. Following screening and baseline assessments (including clinical chemistry, complete blood count, lipid panel, vital signs, and body composition via bioimpedance analysis), eligible participants will be randomly assigned to one of three groups:

1. Amylopectin-chromium blend, 2 g co-ingested with 20 g of protein from yogurt,
2. Amylopectin-chromium blend, 100 mg, co-ingested with 20 g of protein from yogurt, or
3. Placebo (2 g amylopectin) co-ingested with 20 g of protein from yogurt.

Each participant will receive only one product dose during the study. Group assignment will be randomized and blinded to both participants and investigators.

Prior to dosing, participants will undergo exercise familiarization and 5-repetition-maximum testing for leg press and leg extensions. At Visit 3 (Day 5), participants will ingest a single oral dose of ¹⁵N-alanine (2 g) as a metabolic tracer, and then will perform a standardized resistance exercise protocol (3 × 12-15 repetitions each of leg press and leg extension at 60-65 % of estimated 1RM, with 2-minute rest intervals). Immediately following exercise, the assigned study product with yogurt protein will be ingested. A second 20 g yogurt protein serving will be consumed with the evening meal to maintain uniform post-exercise protein intake.

Urinary nitrogen enrichment (¹⁵N-urea) will be measured from 24-hour urine collections (0-12 h and 12-24 h) to determine protein turnover rates. Blood samples obtained at multiple time points will assess biochemical responses, including blood urea nitrogen and isotope enrichment. Whole-body protein synthesis and breakdown will be calculated from tracer kinetics. Continuous glucose monitoring will capture interstitial glucose fluctuations.

Throughout the study, participants will follow a controlled diet standardized for energy and macronutrient content (approximately 1.1 g protein/kg body weight/day) and will abstain from alcohol, caffeine, and strenuous exercise for 24 hours before each visit. Compliance with dietary controls will be verified using the ASA24 or USDA Food Data Central tools.

Adverse events, vital signs, and anthropometrics will be monitored at each visit. The total blood volume collected will be approximately 38 mL. No major safety risks are anticipated; potential discomforts include mild gastrointestinal upset, muscle soreness from resistance exercise, and transient local effects from blood draws.

The primary study outcomes are changes in whole-body protein synthesis and breakdown measured by ¹⁵N-alanine tracer methodology. Secondary outcomes include indices of glucose control, derived from continuous glucose monitoring, and safety/tolerability endpoints.

This study will provide mechanistic insight into the acute effects of the amylopectin-chromium blend on whole-body protein balance in peri- and post-menopausal women, contributing to the broader understanding of nutritional interventions that support muscle health and metabolic function during midlife.

ELIGIBILITY:
Inclusion Criteria:•

Women aged 40-65 years who meet either of the following menstrual-history criteria:

* ≥ 60 days but < 12 months of amenorrhea (late perimenopause)
* Women with ≥ 12 months of spontaneous amenorrhea (post-menopausal)

  * No more than 3 days per week of structured physical activity
  * Provide voluntary signed and dated informed consent.
  * Be in good health and able to participate in an exercise bout as determined by assessment, medical history, and routine blood chemistries.
  * Between the of 40 and 65 years of age (inclusive).
  * Body Mass Index of 18.5-34.9 (inclusive).
  * Body weight of at least 110 pounds.
  * Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5-minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
  * Normal supine, resting heart rate (<90 per minute).
  * Subject agrees to follow standardized controlled diet for 3 days and maintain existing dietary patterns on other days throughout the study period.
  * Subject is willing and able to comply with the study protocol.
  * Able to provide an adequate blood draw.
  * If a dietary supplement was initiated within the past month, the participant is willing to discontinue supplement use followed by a 2-week washout prior to participation in the study. Note: A generic multivitamin is allowed.
  * Refrain from caffeine, exercise, and alcohol for 24 hours prior, and fast for 10 hours prior to each visit.

Exclusion Criteria:

* Current use of any dietary ingredient that impacts glucose control or insulin sensitivity.
* Current vegans or vegetarians.
* Intolerance to dairy foods/drinks.
* Smokes more than 10 cigarettes per day or uses other nicotine products (i.e. vape, patch) that deliver a similar amount of nicotine.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband, etc.).
* Individuals using any kind of GLP-1 medications.
* Other known gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism, e.g. electrolyte abnormalities, diabetes, thyroid disease, adrenal disease, hypogonadism, short bowel syndrome, diarrheal illnesses, history of colon resection, gastric ulcer, reflux disease, gastroparesis, Inborn-Errors-of-Metabolism (such as PKU).
* Individuals who have gained or lost more than 10 pounds within the last 30 days.
* Individuals who are cognitively impaired and/or who are unable to give informed consent.
* Chronic medically diagnosed inflammatory condition or disease (e.g. rheumatoid arthritis, Crohn's disease, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* Medical history of hepatorenal, musculoskeletal, autoimmune, or neurologic disease.
* Known sensitivity to any ingredient in the test formulations as listed in the Certificates-of-Analysis.
* Any other diseases or conditions that, in the opinion of the medical staff, could confound the primary endpoint or place the subject at increased risk of harm if they were to participate.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Whole-Body Protein Turnover (Protein Synthesis and Breakdown) | 24 hours
  This study will evaluate the effect of a dietary supplement consumed with protein and resistance exercise on whole-body protein turnover in healthy adults. Whole-body protein synthesis and breakdown will be assessed using a stable isotope tracer methodology following ingestion of a non-radioactive, isotope-labeled amino acid. Urine and blood samples will be collected over a 24-hour period to quantify protein turnover in response to the intervention.

SECONDARY OUTCOMES:
Interstitial Glucose Concentration measured using 24-24-hour continuous glucose monitoring | Day 0 to day 6
  Interstitial glucose concentrations will be measured continuously using a blinded continuous glucose monitoring system worn on the upper arm. Glucose data will be collected over a 6-day monitoring period and used to derive summary measures including mean glucose concentration and indices of glycemic variability, pre- and post-intervetion

OTHER OUTCOMES:
Blood pressure (systolic and diastolic) | Day 0, 5, and 6
  Systolic and diastolic blood pressure will be measured using a standard automated blood pressure device under resting conditions.
Heart rate | Day 0, 5, and 6
  Heart rate will be measured using a standard automated blood pressure device under resting conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Ziegenfuss, PhD, Principal Investigator — The Center for Applied Health Sciences
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: No